CLINICAL TRIAL: NCT06204809
Title: A Phase 1 Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single-Ascending Doses of PGN-EDODM1 in Adult Participants With Myotonic Dystrophy Type 1 (FREEDOM-DM1)
Brief Title: Safety, Tolerability, PK, and PD Study of PGN-EDODM1 in Participants With Myotonic Dystrophy Type 1
Acronym: FREEDOM-DM1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PepGen Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGN-EDODM1-101
Record Dates: First submitted 2023-12-05; First posted 2024-01-12 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Myotonic Dystrophy 1
Keywords: Myotonic Dystrophy; Muscular Dystrophies; Genetic Diseases, Inborn; Neuromuscular Diseases; Nervous System Diseases; Musculoskeletal Diseases; Myotonic Disorders; Muscular Disorders, Atrophic; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Muscular Diseases; Steinert Disease
MeSH Terms: conditions — Myotonic Dystrophy; Muscular Dystrophies; Genetic Diseases, Inborn; Neuromuscular Diseases; Nervous System Diseases; Musculoskeletal Diseases; Myotonic Disorders; Muscular Disorders, Atrophic; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Muscular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PGN-EDODM1 (Experimental): PGN-EDODM1 for infusion
  Interventions: Drug: PGN-EDODM1 for infusion
- Placebo (Placebo Comparator): 0.9% NaCl
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PGN-EDODM1 for infusion — Single dose of PGN-EDODM1 by intravenous (IV) infusion
  Arms: PGN-EDODM1
Other: Placebo — Administered by IV infusion
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to evaluate the safety and tolerability of single intravenous (IV) doses of PGN-EDODM1 administered to participants with Myotonic Dystrophy Type 1 (DM1).

The study consists of 2 periods: A Screening Period (up to 30 days) and a Treatment and Observation Period (16 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of DM1, as defined as having a repeat sequence in the DMPK gene with at least 100 CTG repeats
* Medical Research Council (MRC) score of ≥ Grade 4- in bilateral tibialis anterior (TA) muscles (the ability to move through full range of motion and hold against at least moderate pressure from the examiner)
* Presence of myotonia

Exclusion Criteria:

* Congenital DM1
* Known history or presence of any clinically significant conditions that may interfere with study safety assessments
* Abnormal laboratory tests at screening
* Medications specific for the treatment of myotonia within 2 weeks prior to screening
* Percent predicted forced vital capacity (FVC) <40%

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events, Serious Adverse Events, with abnormal Clinical Laboratory tests, abnormal ECGs, and abnormal Vital Signs | Baseline to Week 16

SECONDARY OUTCOMES:
Maximum Observed Plasma Drug Concentration (Cmax) of PGN-EDODM1 | Baseline up to Day 3
Time to Maximum Observed Plasma Drug Concentration (Tmax) of PGN-EDODM1 | Baseline up to Day 3
Apparent Terminal Half-Life (t½) of PGN-EDODM1 | Baseline up to Day 3
Area Under the Concentration-time Curve of PGN-EDODM1 | Baseline up to Day 3

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - UCI Center for Clinical Research, Irvine, California
  - Stanford University, Palo Alto, California
  - Rare Disease Research, Atlanta, Georgia
  - University of Kansas Medical Center, Fairway, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - Ottawa Hospital Research Institute (OHRI), Ottawa, Ontario
  - CIUSSS du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
- United Kingdom (2):
  - University College London Hospital, London, UK
  - Salford Royal Hospital, Salford